CLINICAL TRIAL: NCT07213323
Title: Evaluation of the Efficacy of Probiotics on Digestive Quality of Life in Patients Initiating GLP-1 Receptor Agonists for the Treatment of Obesity. A Randomized, Double-blind Trial
Brief Title: Probiotic Intervention for Digestive Health in Obese Patients Initiating GLP-RA Treatment
Acronym: PROBIO-GLP1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 69HCL25_0321; 2025-A01248-41 (Other: ID-RCB)
Record Dates: First submitted 2025-09-18; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obesity &Amp; Overweight; Digestive Disorders
Keywords: GLP1 R-agonist; Probiotics; Quality of life
MeSH Terms: conditions — Obesity; Overweight; Digestive System Diseases | interventions — Probiotics; Biological Products

STUDY DESIGN:
Intervention Model Description: Prospective, double blind, randomized, monocentric, 2 parallel groups (1:1) study evaluating superiority probiotics over placebo in limiting the impairment in digestive quality of life over 24-week in patients with obesity initiating GLP-1 RA (semaglutide or tirzepatide) for weight control.
Who Masked: Participant, Investigator
Masking Description: Double-blind study : patients and investigators will not be informed of the approach (probiotics or placebo ) which will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Obese subjects who are going to start a GLP-1 R-agonist (semaglutide or tirzepatide) as part of their weight management in routine clinical practice will received during 26 weeks 1 capsule a day every morning of probiotics that will begin 2 weeks before the initiation of semaglutide or tirzepatide treatment.
  Interventions: Dietary Supplement: Probiotics (Natural product)
- Placebo (Placebo Comparator): Obese subjects who are going to start a GLP-1 R-agonist (semaglutide or tirzepatide) as part of their weight management in routine clinical practice will received during 26 weeks 1 capsule a day every morning of PLACEBO that will begin 2 weeks before the initiation of semaglutide or tirzepatide treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics (Natural product) — Participants will be instructed to daily take, during 26 weeks (that will begin 2 weeks before the initiation of semaglutide or tirzepatide treatment) one capsule of a probiotic with water at room temperature with the first meal.
  Dosage levels: 1 capsule Digestive Quality of life during the study will be assessed.
  Arms: Probiotics
Other: Placebo — Participants will be instructed to daily take, during 26 weeks (that will begin 2 weeks before the initiation of semaglutide or tirzepatide treatment) one capsule of PLACEBO with water at room temperature with the first meal.
  Digestive Quality of life during the study will be assessed.
  Arms: Placebo

SUMMARY:
Obesity is a prevalent chronic disease affecting 17% of the French population. Treatment involves multiple factors, with pharmacotherapy playing an increasingly important role. GLP-1 receptor agonists (GLP1 RAs) are considered revolutionary in obesity treatment, with three approved molecules available in France: liraglutide, semaglutide, and tirzepatide. These treatments, combined with a healthy lifestyle, induce significant weight loss: 9% with liraglutide, 15% with semaglutide, and 20% with tirzepatide.

The most common adverse events (AEs) associated with GLP-1 RAs are gastrointestinal (GI) disorders, including nausea, vomiting, diarrhea, and abdominal pain. These AEs are dose-dependent and often decline over time. In phase 3 trials, semaglutide 2.4 mg showed higher rates of GI AEs compared to placebo, but most were mild to moderate and transient. GI AEs led to dose reduction or temporary treatment interruption in 12.5% of participants, with few permanent discontinuations.

Probiotics, are live microorganisms that benefit the host by improving gut microflora. Probiotics has been clinically proven to benefit gastrointestinal health. Probiotics may reduces symptoms of irritable bowel syndrome (IBS), improves gut barrier function, reduces inflammation, and decreases the incidence of C. difficile infection (CDI) in patients taking antibiotics.

Probiotics is therefore theorized to potentially reduce GI side effects associated with GLP-1 RA treatment for obesity.

Hypothesis Probiotics will prevent and limit the digestive disorders induced by GLP-1 R agonists, particularly during the dose escalation period. This would allow better digestive tolerance of the treatments, limiting the number of definitive treatment interruptions, facilitating compliance and dose escalation with a larger number of subjects at full dose and therefore with better systemic exposure to the compounds, a key factor in their effects on weight loss.

DETAILED DESCRIPTION:
Obesity is a prevalent chronic disease affecting 17% of the French population. Treatment involves multiple factors, with pharmacotherapy playing an increasingly important role. GLP-1 receptor agonists (GLP1 RAs) are considered revolutionary in obesity treatment, with three approved molecules available in France: liraglutide, semaglutide, and tirzepatide. These treatments, combined with a healthy lifestyle, induce significant weight loss: 9% with liraglutide, 15% with semaglutide, and 20% with tirzepatide.

The most common adverse events (AEs) associated with GLP-1 RAs are gastrointestinal (GI) disorders, including nausea, vomiting, diarrhea, and abdominal pain. These AEs are dose-dependent and often decline over time. In phase 3 trials, semaglutide 2.4 mg showed higher rates of GI AEs compared to placebo, but most were mild to moderate and transient. GI AEs led to dose reduction or temporary treatment interruption in 12.5% of participants, with few permanent discontinuations.

Probiotics, are live microorganisms that benefit the host by improving gut microflora. Probiotics has been clinically proven to benefit gastrointestinal health. Probiotics may reduces symptoms of irritable bowel syndrome (IBS), improves gut barrier function, reduces inflammation, and decreases the incidence of C. difficile infection (CDI) in patients taking antibiotics.

Probiotics is therefore theorized to potentially reduce GI side effects associated with GLP-1 RA treatment for obesity.

Hypothesis Probiotics will prevent and limit the digestive disorders induced by GLP-1 R agonists, particularly during the dose escalation period. This would allow better digestive tolerance of the treatments, limiting the number of definitive treatment interruptions, facilitating compliance and dose escalation with a larger number of subjects at full dose and therefore with better systemic exposure to the compounds, a key factor in their effects on weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is going to start a GLP-1 RA (semaglutide or tirzepatide) for weight management
* Men or Women
* BMI ≥ 30 kg/m2 or BMI ≥ 27 kg/m2 associated with one or more co-morbidities (arterial hypertension, sleep apnea, dyslipidemia, arthritis)
* Between 18 and 75 years old
* In the opinion of the investigator, the patient must have adequate support to comply with the entire study requirements as described in the protocol (e.g. transportation to and from trial site, ability to understand and fill the self-rating scales, drug compliance, availability to attend to the scheduled visits, etc…).
* Patient who agrees to be included in the study and who signs the informed consent form
* Female participants of childbearing potential must agree to use effective contraception
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

Criteria relating to the study population:

* Patients under 18 years old
* Patient with contraindication to semaglutide or tirzepatide according to the Summary of Product Characteristics (SPC).
* Patients scheduled for bariatric surgery during the study period
* Patients who have had bariatric surgery in the last 12 months
* Patient with a current diagnosis of diabetes.
* Patients with a current diagnosis of liver cirrhosis, short bowel syndrome or inflammatory bowel disease (IBD).
* Patients with severely weakened immune system.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine, or other systemic disease.

Product criteria:

Patient with known allergy to the product of the study

Prohibited treatments :

Current associated treatments or used in the last 30 days: GLP-1 RA, Anti-obesity drugs (AOD), Corticosteroids, Atypical neuroleptics, Antibiotics, Probiotics, Prebiotics

Regulatory criteria :

* Persons deprived of their liberty by a judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Subjects participating in other interventional research with an exclusion period still in progress at pre-inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Limitation of the impairment in digestive quality of life during the dose escalation of GLP1-RA (semaglutide or tirzepatide) | Every 5 weeks
  Assessment using partial GIQLI Score (5 items: 1,27,31,32,33 of the total GIQLI) in each GLP-1 RA group measured 4 weeks following the previous dose escalation, with the GLP1-RA dose standardized on a 0-1 scale.
  Item 1 for abdominal pain, Item 27 for dyspepsia, Item 31 for diarrhea, item 32 for constipation and Item 33 for nausea.
  For each item, 5 responses will be proposed to the patients and for each answer, a score ranging from 0 to 4 will be assigned The highest score is 20 and defines a more favorable health state

SECONDARY OUTCOMES:
Digestive quality of life | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison between the probiotic group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of the partial GIQLI Scores (Questions 1,27,31,32,33). Item 1 for abdominal pain, Item 27 for dyspepsia, Item 31 for diarrhea, item 32 for constipation and Item 33 for nausea.
  For each item, 5 responses and for each answer, a score ranging from 0 to 4. The highest score is 20 and defines a more favorable health state
Nausea | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison of nausea between the probiotic group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of partial GIQLI score (question 33) of nausea score ranging from 0 to 4.
  4 defines the more favourable score
Dyspepsia | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison of dyspepsia between the probiotic group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of partial GIQLI score (question 27) of dyspepsia score ranging from 0 to 4.
  4 defines the more favourable score
Diarrhea | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison of diarrhea between the probiotics group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of partial GIQLI score (question 31) of diarrhea score ranging from 0 to 4.
  4 defines the more favourable score
Constipation | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison of constipation between the probiotic group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of partial GIQLI score (question 32) of constipation score ranging from 0 to 4.
  4 defines the more favourable score
Abdominal pain | From baseline to 4, 8, 12, 16, 20 and 24 weeks of treatment
  Comparison of abdominal pain between the probiotic group and placebo group in the whole population and in the subpopulation of subjects having reached the planned GLP-1 RA treatment dose at 24 weeks, according to the dose escalation design:
  Evolution of partial GIQLI score (question 1) of abdominal pain score ranging from 0 to 4.
  4 defines the more favourable score
GLP-1 receptor agonist dosage | 4, 8, 12, 16, 20 and 24 weeks of intervention
  Average GLP-1 RA dose
GLP1-RA dose escalation | 4, 8, 12, 16, 20 and 24 weeks of intervention
  Proportion of patients having reached the planned GLP-1 RA treatment dose according to the dose escalation protocol at 4, 8, 12, 16, 20 and 24 weeks
GLP1-RA dose discontinuation/maintenance | 4, 8, 12, 16, 20 and 24 weeks of intervention
  Proportion of patients who had to reduce or to interrupt definitively their GLP-1 RA treatment dose at 4, 8, 12, 16, 20 and 24 weeks
Weight loss | 4, 8, 12, 16, 20 and 24 weeks of intervention
  Percent of weight change from baseline
Weight loss | 4, 8, 12, 16, 20 and 24 weeks of intervention
  absolute change in body weight from baseline
Weight loss | 4, 8, 12, 16, 20 and 24 weeks of intervention
  Rate of patients achieving a body weight reduction of ≥5%, ≥10%, ≥15%
Quality of life assessed with GIQLI questionnaire | baseline, 12 and 24 weeks of treatment
  This questionnaire consists of 36 items exploring 5 dimensions or subscales: symptoms, physical condition, emotions, social integration and the effect of any medical treatment. For each item, 5 responses will be proposed to the patients and for each answer, a score ranging from 0 to 4 (highest score = 144) will be assigned. A high score defines a more favorable health state.
Quality of life assessed with SF36 questionnaire | baseline, 12 and 24 weeks of treatment
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/tiredness, and general health perceptions. It also includes a single item that provides an indication of a perceived change in health
Fat mass | Baseline, before implementation of GLP1-RA, 12 and 24 weeks of treatment
  Measurement of fat mass will explore the body composition. Results will be expressed in kg and %
Lean mass | Baseline, before implementation of GLP1-RA, 12 and 24 weeks of treatment
  Measurement of lean mass will explore the body composition. Results will be expressed in kg and %
Skeletal muscle mass | Baseline, before implementation of GLP1-RA, 12 and 24 weeks of treatment
  Measurement of skeletal muscle mass will explore the body composition. Results will be expressed in kg and %
Adverse Events | After 4, 8, 12, 16, 20 and 24 weeks of treatment.
  The safety will be assessed by the Number of adverse events, linked or not to the study product
Severe Adverse Events | After 4, 8, 12, 16, 20 and 24 weeks of treatment.
  The safety will be assessed by the number of severe adverse events, linked or not to the study product
Intestinal microbiota | Baseline and 24 weeks of treatment
  Fecal microbiota composition

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, PUPH, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France